CLINICAL TRIAL: NCT06973551
Title: The Benefits of Nostalgia-Based Virtual Reality Brain Health Interventions on Nostalgia Tendencies, Life Satisfaction, Psychological Well-Being, Depression Levels, and Cognitive Function in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202503HM026
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia; Cognitive Decline; Psychological Well-being
Keywords: Older adults; Mild Cognitive Impairment; Dementia; Cognitive Training; nostalgia-based virtual reality; Aging and Cognitive Health; Virtual Reality Cognitive Training
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel-group randomized controlled trial design. Eligible participants are randomly assigned to either an experimental group (receiving nostalgia-based VR cognitive training) or a control group (engaging in routine weekly activities without specific intervention). The study period spans 12 weeks, enabling direct comparison of outcomes between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nostalgia-Based VR Cognitive Training (Experimental): Participants in this arm will receive the "Brain Health Nostalgic VR Program," a culturally grounded virtual reality intervention integrating nostalgic elements representative of Taiwanese culture (e.g., old photographs, household objects, traditional media, and familiar scenarios) with interactive cognitive training. The training targets seven domains: attention, imagination and creativity, observation, memory, reasoning, reading comprehension, and thinking. Each weekly session spans 60-90 minutes in total, including setup, support, and breaks, while the actual VR usage time is 10-30 minutes depending on individual tolerance. The intervention is conducted weekly over 12 weeks at the participant's care facility, with full assistance and monitoring by the research team.
  Interventions: Behavioral: Brain Health Nostalgic VR Program
- Routine Weekly Activities (No Intervention): Participants in this arm will continue with their routine weekly activities provided by their respective long-term care facilities. These activities may include light physical exercise, social engagement, passive entertainment (e.g., watching TV), or unstructured leisure. No structured cognitive training or VR-related content will be administered. This arm serves as a control group for comparison with the experimental group receiving the nostalgia-based VR intervention.

INTERVENTIONS:
Behavioral: Brain Health Nostalgic VR Program — The "Brain Health Nostalgic VR Program" is a culturally tailored virtual reality intervention integrating nostalgic content from Taiwanese culture (e.g., vintage photographs, familiar objects, historical TV clips, traditional settings) with interactive cognitive training tasks. The program targets seven cognitive domains: attention, imagination and creativity, observation, memory, reasoning, reading comprehension, and thinking. Each weekly session spans 60-90 minutes, with 10-30 minutes of actual VR use based on participant tolerance, each participant will use VR for no more than 30 minutes per session before taking a break. The intervention is delivered once per week over a 12-week period in long-term care settings, with researcher support provided throughout.
  Other Names: nostalgia-based virtual reality; Elderly Brain Boosting Nostalgic VR; Nostalgia-Based VR Cognitive Training
  Arms: Nostalgia-Based VR Cognitive Training

SUMMARY:
This randomized controlled trial investigates the effects of a nostalgia-based cognitive training intervention delivered via Virtual Reality (VR) on emotional well-being and cognitive functioning among community-dwelling older adults (≥65 years) in northern Taiwan, specifically targeting those with mild cognitive impairment (MCI) or mild dementia. The study, conducted at National Taiwan Normal University, aims to assess whether engaging older adults in nostalgic VR experiences can enhance nostalgia proneness, life satisfaction, and psychological well-being, while also reducing depressive symptoms and improving cognitive functions.

Participants who meet inclusion criteria (aged 65+, capable of communicating in Mandarin or Taiwanese, without severe psychiatric conditions, with sufficient vision/hearing) will be randomly assigned to either the experimental group receiving the "Brain Health Nostalgic VR Program" or a control group engaged in routine weekly activities. Each weekly session spans 60-90 minutes in total, including setup, support, and breaks, while the actual VR usage time is 10-30 minutes depending on individual tolerance. Research staff will provide close support and safety monitoring during all sessions.

Pre- and post-intervention outcomes will be measured using standardized assessments: Southampton Nostalgia Scale (SNS), Short-Form Life Satisfaction Index (LSI-SF), Geriatric Depression Scale (GDS-15), Short-Form Chinese version of Ryff's Psychological Well-being Scale (PWB-18), and the Montreal Cognitive Assessment Taiwan Version (MoCA-T). The study emphasizes participant safety and data confidentiality throughout its duration. Findings aim to demonstrate VR's potential as a non-invasive, preventive strategy for cognitive decline and mental health enhancement among older populations.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) examines the effectiveness of a culturally tailored, nostalgia-based virtual reality (VR) program in promoting cognitive health and emotional well-being among older adults (≥65 years) in northern Taiwan. The study is designed in response to Taiwan's rapid transition into a super-aged society, where dementia prevalence and caregiving burdens are expected to rise significantly. Mild cognitive impairment (MCI) represents a critical transitional state with cognitive plasticity, providing a valuable opportunity for early non-pharmacological intervention.

Theoretical Framework

The intervention is guided by Expectation Confirmation Theory (ECT), which emphasizes how perceptions of usefulness, ease of use, and enjoyment influence participants' satisfaction and long-term intention to adopt health-related technologies. This framework allows the study to move beyond clinical outcomes and assess the feasibility and sustainability of VR interventions among older adults.

Intervention Features

The Brain Health Nostalgic VR Program integrates reminiscence therapy with cognitive training within immersive VR. The content is uniquely designed with Taiwan-specific cultural elements, such as traditional wedding rituals, historical films, and familiar objects from everyday life, to evoke strong nostalgic responses and enhance emotional engagement.

Cognitive exercises are embedded in the VR environment and target seven domains:Attention, Memory, Reasoning, Reading comprehension, Thinking skills, Imagination and creativity, Observational skills.

Each weekly session lasts approximately 60-90 minutes, including preparation, VR exposure (10-30 minutes depending on tolerance), discussion, and breaks. The intervention continues for 12 times, with both short-term (8-12 weeks) and longer-term (24 weeks) follow-up assessments. Sessions are delivered within participants' own care facilities to ensure safety and comfort.

Distinguishing Characteristics

Unlike conventional reminiscence therapy, which often uses photos or group conversations, the immersive VR environment minimizes external distractions and enhances the sense of presence. This approach is expected to amplify the therapeutic benefits of reminiscence by combining emotional stimulation with structured cognitive tasks.

Previous studies in Asia and Europe have shown promising results from VR-based reminiscence and cognitive training, but most were limited by small sample sizes or short-term pilot designs. This trial is one of the first large-scale, culturally adapted RCTs in Taiwan, addressing both psychological outcomes (e.g., life satisfaction, well-being, depressive symptoms) and cognitive performance in older adults with MCI or mild dementia.

Anticipated Contributions

This study aims to:

Demonstrate the efficacy of a VR-based nostalgia and cognitive training program as an innovative non-pharmacological intervention.

Provide empirical evidence on how culturally tailored VR content can enhance reminiscence, reduce depressive symptoms, and improve cognitive functioning in older adults.

Evaluate user acceptance and long-term adoption intentions, offering insights into the scalability of digital health interventions in community and institutional settings.

By integrating cultural reminiscence, cognitive stimulation, and immersive VR technology, this trial contributes to both the scientific evidence base and practical strategies for dementia prevention, elderly mental health promotion, and caregiver burden reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Able to communicate in Mandarin or Taiwanese
* Capable of wearing and operating a VR headset and handheld controllers
* Sufficient vision and hearing to interact with VR content (assistive devices permitted)
* Able to provide informed consent or have a legal guardian provide consent

Exclusion Criteria:

* Diagnosis of severe dementia or advanced neurodegenerative disease
* Severe psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Major visual or auditory impairments that would interfere with VR use, even with assistive devices
* Unconsciousness, inability to stay awake or focused for the session duration Inability to comply with study protocol or scheduled sessions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function Assessed by MoCA-T | Baseline, Week 12, Week 24
  Cognitive function will be measured using the Montreal Cognitive Assessment - Taiwan Version (MoCA-T), a validated tool for detecting mild cognitive impairment (MCI) and early dementia. The MoCA-T assesses multiple domains including memory, attention, executive function, language, and visuospatial skills.
  Score range: 0-30 Interpretation: Higher scores indicate better cognitive functioning. For the Taiwanese version, a cutoff score of 23/24 has been suggested as the optimal threshold for distinguishing MCI patients from cognitively normal controls.

SECONDARY OUTCOMES:
Change in Nostalgia Proneness Assessed by Southampton Nostalgia Scale (SNS) | Baseline, Week 12, Week 24
  Change in Nostalgia Proneness Assessed by the Southampton Nostalgia Scale (SNS) Nostalgia proneness will be measured using the 7-item Southampton Nostalgia Scale (SNS), which evaluates both the importance/meaning of nostalgia (items 1-4) and the frequency of nostalgic experiences (items 5-7). Items 1-6 are rated on a 7-point Likert scale (1-7). Importance items range from 1 = not at all valuable/important to 7 = very valuable/important. General frequency items range from 1 = very rare to 7 = very frequent. Item 7 specifically assesses the concrete frequency of nostalgic experiences with options ranging from 1 = once or twice a year to 7 = at least once a day. The total score ranges from 7 to 49, with higher scores indicating a stronger proneness to nostalgia.
Change in Depression Symptoms Assessed by GDS-15 | Baseline, Week 12, Week 24
  Depression levels will be measured using the 15-item Geriatric Depression Scale (GDS-15), a validated self-report tool for older adults. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms. The measure will be administered at baseline, week 12, and week 24.
Change in Psychological Well-being Assessed by PWB-18 | Baseline, Week 12, Week 24
  Psychological well-being will be evaluated using the 18-item Short-Form Chinese version of Ryff's Psychological Well-being Scale (PWB-18), which measures six dimensions of well-being. Higher scores indicate greater psychological well-being. The scale will be administered at baseline, week 12, and week 24.
Change in Life Satisfaction Assessed by LSI-SF | Baseline, Week 12, Week 24
  Change in Life Satisfaction Assessed by the Life Satisfaction Index - Short Form (LSI-SF) Life satisfaction will be assessed using the 6-item Life Satisfaction Index - Short Form (LSI-SF), derived from the original Life Satisfaction Index-A (LSIA) by Neugarten et al. (1961). The items cover three domains: (1) zest vs. apathy, (2) resolution and fortitude, and (3) congruence between desired and achieved goals. One item ("Most of the things I do are boring or monotonous") is reverse-coded. Each item is scored dichotomously (0 = no, 1 = yes), yielding a total score ranging from 0 to 6. Higher scores indicate greater life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Long Guo, PhD, Study Chair — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available after publication of the main trial results in an international peer-reviewed journal. Access requires a formal request to the corresponding author and approval. Shared data will include variables related to primary and secondary outcomes (e.g., demographics, cognitive function, well-being, depression, and life satisfaction). Data will be provided for academic, non-commercial research only, beginning 6 months after publication and up to 3 years thereafter. Qualified researchers must submit a sound proposal; upon approval, data will be securely transferred electronically.